CLINICAL TRIAL: NCT06622759
Title: The Use of a Porcine Collagen Matrix for the Prevention of Buccal Bone Wall During Implant Placement in the Aesthetic Zone. A Randomized Controlled Clinical Trial.
Brief Title: The Use of a Porcine Collagen Matrix for the Prevention of Buccal Bone Wall Resorption During Implant Placement in the Aesthetic Zone.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Ioannis Vouros, Study Chair: Ioannis Vouros, DDS, PhD, Professor of Periodontology, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20/29-06-2023
Record Dates: First submitted 2024-09-13; First posted 2024-10-02 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Soft Tissue Augmentation
Keywords: Implants; Esthetic zone; Soft tissue augmentation; Collagen matrix; Soft tissue grafts; Connetive Tissue Graft; Porcine collagen matrix
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- No Graft (Other): In the control group, the implant will be placed without any kind of soft tissue graft. Also, it will be placed at the level of the bone and the flaps will be sutured with 5/0 absorbable sutures.
  Interventions: Procedure: Control group
- CTG (Experimental): In the first experimental group, prosthetically guided implant placement will be performed as well as an increase of the soft tissue volume with an autologous Connective Tissue Graft (CTG). The implant will be placed up to the level of the bone. The autologous graft will be harvested either from the palate as a free gingival graft or as a subepithelial graft, or from the maxillary cusps. The graft will be immobilized in the buccal flap with two simple interrupted sutures and 5/0 absorbable sutures covering the buccal and coronal surfaces of the alveoral bone. Finally, the flap will be displaced coronally so that we have closure in the first place.
  Interventions: Procedure: CTG
- Collagen Matrix (Experimental): In the second experimental group, prosthetically guided implant placement and simultaneous soft tissue volume augmentation with porcine Collagen Matrix (CM) - Geistlich FibroGide - will be performed. Initially, full-thickness flap will be raised mainly buccally but also palatally. The implant will then be placed at the level of the bone. The flap will buccally become partial thickness and full thickness again so that we can move it coronally to cover and perfuse the graft. The collagenous graft will be shaped to fit the surgical site, be covered by the periosteum, and will completely cover the buccal bone. Also, it should expand coronal to the alveoral crest. Two horizontal matress sutures (P.G.A 5/0 absorbable) will immobilize the graft. Finally, the buccal flap will be displaced coronally, so that we have convergence in the first place.
  Interventions: Procedure: Collagen Matrix

INTERVENTIONS:
Procedure: CTG — Connective Tissue Graft has been widely used around implants to increase either the thickness of the soft tissues or the width of keratinized tissues. It is considered the gold standard for soft tissue grafting. The main drawbacks are the donor morbidity and the limit amount of intraoral donor sites. In this study it will be used in the test 1 group in order to compare its clinical results with the other groups.
  Arms: CTG
Procedure: Collagen Matrix — Collagen matrix has been used in several studies in order to evaluate its clinical properties over the last years. In this study, the graft will be placed buccally at the time of implant placement in the aesthetic zone in order to assess its clinical and radiographic properties in terms of buccal bone resorption and soft tissue augmentation. Histological assessment and Patient Reported outcomes will also be evaluated.
  Arms: Collagen Matrix
Procedure: Control group — In the control group, the implant will be placed without any kind of soft tissue graft in order to compare this treatment modality that many clinicians apply at the clinical practice.
  Arms: No Graft

SUMMARY:
Aim:

To provide a comparative assessment of the clinical and radiographic effect of porcine collagen matrix when placed buccally at the time of single implant placement in the aesthetic zone vs autogenous connective tissue graft in terms of buccal bone resorption and soft tissue augmentation 6 months post operative. Histological assessment and patient reported outcomes were reported

DETAILED DESCRIPTION:
Introduction: The need to restore lost teeth with dental implants is now a daily practice. In particular, treatments aimed at replacing lost teeth in the upper anterior aesthetic zone are particularly demanding, in terms of evaluating functional and aesthetic factors that influence the result. In order to successfully maintain the implants in the long term and to ensure aesthetics, there must be adequate dimensions of the alveolar crest and especially a satisfactory range of buccal bone in the area of placement. There are reports, that in areas with reduced width and thickness of soft tissues, there is a risk of resorption and further loss of buccal plate after implant placement which can lead to deterioration of aesthetics. For this reason soft tissue augmentation using soft tissue grafts may lead to a decrease in buccal bone resorption. According to the above, it would be of particular interest to investigate the possibility of using a material such as the collagen matrix as an alternative procedure for soft tissue augmentation, compared to the conventional use of a subepithelial connective tissue graft, which is associated with greater morbidity and complicates the surgical procedure.

So, the investigators designed a prospective, randomized controlled clinical trial of 6 months duration. The 36 participants will be periodontally healthy or periodontally treated patients, who seek treatment at the clinic of Periodontology and Implantology of the Department of Dentistry, Aristotle University Thessaloniki.The participants should have completed Step 1 and 2 of periodontal treatment at least 3 months before being enrolled. If periodontally healthy, they will have received a session of supragingival removal of deposits and they will be given oral hygiene instructions. Patients should need implant reconsruction in the upper anterior esthetic zone without need for a prior bone augmentation procedure to increase the dimensions of the bone substrate. After the initial clinical evaluation for the appropriateness of the case, a consent form will be signed by the participants and then the patients will be randomized to one of the three treatment groups.In the control group, 12 patients will undergo prosthetically guided implant placement without increasing soft tissue volume. In the first experimental group, the next 12 patients will receive prosthetically guided implant placement and simultaneous volume increase of the soft tissues with a collagenous matrix of porcine origin (Geistlich Fibro-Gide), while in the second experimental group (12 patients), the volume increase of the soft tissues will be performed with a subepithelial connective tissue graft from the palate.The evaluation of the therapeutic outcome will be based on (a) clinical parameters (bleeding on probing, plaque index, extent of keratinized gingiva), (b) measurement of soft tissue thickness with an ultrasound device (Pirop Ophthalmic Scanner, Echoson Company, Poland. A scan Probe 20MHz) (c) radiographic parameters (Cone Beam Computed Tomography immediately after dental implant placement and 6 months postoperatively) and (d) histological examination of the soft tissues during the exposure of the implants at 3 months.The tissue biopsy will be taken from the coronal part of the alveolar crest. Finally, the participants will be asked to complete a questionnaire to assess the experience and subjective perception and discomfort after surgical treatment.The re-assesment in 3 months will include exposing the dental implant and taking the tissue for biopsy. Finally, at 6 months postoperatively, the clinical parameters mentioned above will be evaluated, the thickness of the soft tissues will be measured with the ultrasound device and radiographic control with cone beam computed tomography to measure the thickness of the buccal bone plate.

Schedule and clinical procedures for both treatment groups:

First visit- Initial examination at least 3 months after the end of periodontal treatment Medical dental history Patient participation eligibility check - written consent - randomization Taking intraoral photographs Periodontontal chart recording: Pocket depth (PD), Clinical attachment loss (CAL), Bleeding on probing (BoP), Keratinized tissue width (KT), Soft Tissue Thickness (STH) with an ultrasound device, Buccal Bone Thickness (BBT) through bone sounding using a customized splint.

Taking a periapical radiograph in the area of interest with a parallel technique.

Repetition of oral hygiene instructions (Soft toothbrush Modified Bass technique, Interdental cleaning) Removal of supragingival deposits.

Second visit- Baseline Implant placement in experimental or control group. Modification of oral hygiene instructions - Post-operative instructions. Taking intraoral photographs Radiographic examination by Cone Beam Computed Tomography (CBCT)

Third visit (2 weeks after surgery) - Suture removal - Assessment of healing Removal of sutures Healing control Oral hygiene instructions Taking intraoral photographs Completing a questionnaire

Forth visit (3 months after placement of implants) - Second stage procedure the - Taking a piece of tissue for biopsy Surgical exposure of implant Obtain tissue for biopsy Oral hygiene instructions

Fifth visit (6 months after placement of the implants) - Radiographic examination Periodontal chart recording: Pocket depth (PD), Clinical attachment loss (CAL), Bleeding on probing (BoP), Keratinized tissue (KT), Measurement of Soft Tissue Thickness (STH) with ultrasound device and customized splint Radiographic screening by cone beam computed tomography (CBCT) to measure the Buccal Bone Thickness Repeat oral hygiene instructions Taking intraoral photographs

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy adult patients.
2. 18 years or older.
3. Need for replacement of single implant in the upper aesthetic zone (second premolar to second premolar)
4. Ridge width (bucco-lingual) no greater than 6 mm at its narrowest point.
5. Minimum 2mm of attached gingiva.
6. Ability to comply with the study related procedures such as exercising good oral hygiene and attending all follow-up examinations.
7. Ability to fully understand the nature of the proposed surgery and ability to sign the informed consent form

Exclusion Criteria:

1. Poor oral hygiene (FMPS < 20%, FMBS < 15%) and poor motivation
2. Heavy smokers (>10 cigarettes per day)
3. Need for bone augmentation
4. Untreated periodontitis
5. General contraindications for dental and/or surgical treatment
6. History of malignancy, radiotherapy, or chemotherapy for malignancy within the past 5 years
7. Women of child bearing age, not using a standard accepted method for contraception
8. Pregnancy or breast feeding
9. Previous and concurrent medication affecting mucosal healing in general (e.g. steroids, large doses of anti-inflammatory drugs
10. Disease affecting connective tissue metabolism (e.g. collagenases)
11. Allergy to collagen

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2025-08-20 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Soft Tissue Thickness | 6 months
  Thickness of soft tissue buccally
Buccal Bone Thickness | 6 months
  Thickness of marginal bone buccally

SECONDARY OUTCOMES:
Keratinized tissues | 6 months
  Width of keratinized tissues in mid-buccal aspect of implant

OTHER OUTCOMES:
Full Mouth Bleeding Score | 6 months
  Full Mouth Bleeding Score: Percentage of tooth sites with bleeding when a periodontal probe is traced along the gingival margin. Range: 0-100% (the lower the percentage, the better the clinical outcome).
Full mouth plaque score | 6 months
  Full Mouth Plaque Score: Percentage of tooth sites with detectable plaque deposits. Range: 0-100% (the lower the percentage, the better the clinical outcome).
PROMs (Patient Relative Outcome Measures) | 14 days (after surgical treatment)
  Patients will be asked to complete a questionnaire to assess the experience and subjective perception and discomfort immediatelly 10 days after the surgical procedure (during sutures removal).

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Vouros, DDS, Ph.D, Study Chair — Aristotle Univerity of Thessaloniki
Locations (1):
- Department of Preventive Dentistry, Periodontology & Implant Biology, School of Dentistry, Aristotle University, Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Linkevicius T, Apse P, Grybauskas S, Puisys A. Reaction of crestal bone around implants depending on mucosal tissue thickness. A 1-year prospective clinical study. Stomatologija. 2009;11(3):83-91. PMID 19996674
- [Background] Linkevicius T, Apse P, Grybauskas S, Puisys A. The influence of soft tissue thickness on crestal bone changes around implants: a 1-year prospective controlled clinical trial. Int J Oral Maxillofac Implants. 2009 Jul-Aug;24(4):712-9. PMID 19885413
- [Background] Puisys A, Linkevicius T. The influence of mucosal tissue thickening on crestal bone stability around bone-level implants. A prospective controlled clinical trial. Clin Oral Implants Res. 2015 Feb;26(2):123-9. doi: 10.1111/clr.12301. Epub 2013 Dec 9. PMID 24313250
- [Background] Puisys A, Deikuviene J, Vindasiute-Narbute E, Razukevicus D, Zvirblis T, Linkevicius T. Connective tissue graft vs porcine collagen matrix after immediate implant placement in esthetic area: A randomized clinical trial. Clin Implant Dent Relat Res. 2022 Apr;24(2):141-150. doi: 10.1111/cid.13058. Epub 2022 Mar 24. PMID 35324053
- [Background] Thoma DS, Zeltner M, Hilbe M, Hammerle CH, Husler J, Jung RE. Randomized controlled clinical study evaluating effectiveness and safety of a volume-stable collagen matrix compared to autogenous connective tissue grafts for soft tissue augmentation at implant sites. J Clin Periodontol. 2016 Oct;43(10):874-85. doi: 10.1111/jcpe.12588. Epub 2016 Aug 12. PMID 27310522
- [Background] Thoma DS, Gasser TJW, Jung RE, Hammerle CHF. Randomized controlled clinical trial comparing implant sites augmented with a volume-stable collagen matrix or an autogenous connective tissue graft: 3-year data after insertion of reconstructions. J Clin Periodontol. 2020 May;47(5):630-639. doi: 10.1111/jcpe.13271. PMID 32096246
- [Background] Giannobile WV, Jung RE, Schwarz F; Groups of the 2nd Osteology Foundation Consensus Meeting. Evidence-based knowledge on the aesthetics and maintenance of peri-implant soft tissues: Osteology Foundation Consensus Report Part 1-Effects of soft tissue augmentation procedures on the maintenance of peri-implant soft tissue health. Clin Oral Implants Res. 2018 Mar;29 Suppl 15:7-10. doi: 10.1111/clr.13110. PMID 29498127
- [Background] Atieh MA, Alsabeeha NHM. Soft tissue changes after connective tissue grafts around immediately placed and restored dental implants in the esthetic zone: A systematic review and meta-analysis. J Esthet Restor Dent. 2020 Apr;32(3):280-290. doi: 10.1111/jerd.12538. Epub 2019 Nov 4. PMID 32311199
- [Background] Thoma DS, Naenni N, Figuero E, Hammerle CHF, Schwarz F, Jung RE, Sanz-Sanchez I. Effects of soft tissue augmentation procedures on peri-implant health or disease: A systematic review and meta-analysis. Clin Oral Implants Res. 2018 Mar;29 Suppl 15:32-49. doi: 10.1111/clr.13114. PMID 29498129
- [Background] Puzio M, Blaszczyszyn A, Hadzik J, Dominiak M. Ultrasound assessment of soft tissue augmentation around implants in the aesthetic zone using a connective tissue graft and xenogeneic collagen matrix - 1-year randomised follow-up. Ann Anat. 2018 May;217:129-141. doi: 10.1016/j.aanat.2017.11.003. Epub 2017 Dec 15. PMID 29248711
- [Background] Valles C, Vilarrasa J, Barallat L, Pascual A, Nart J. Efficacy of soft tissue augmentation procedures on tissue thickening around dental implants: A systematic review and meta-analysis. Clin Oral Implants Res. 2022 Jun;33 Suppl 23:72-99. doi: 10.1111/clr.13920. PMID 35763023